CLINICAL TRIAL: NCT02961049
Title: Influences of Gingival Cord Retractor in Retention Rate of Non-carious Cervical Lesions Restorations With Different Adhesive Systems. Randomized Clinical Trials.
Brief Title: Influences of Gingival Cord Retractor in Retention Rate of Non-carious Cervical Lesions Restorations.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, PAULO VINICIUS SOARES, Professor, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE - 57032016.0.0000.5152
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Dental Wear; Tooth Wear
MeSH Terms: conditions — Tooth Wear | interventions — Therapeutic Irrigation; Desiccation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Retraction and total-etch (Active Comparator): Gingival displacement with a gingival cord (#0, #00 or #000) prior to the restoration. Application of total-etch adhesive system: enamel and dentin etched with 35% phosphoric acid, wash, dry, two layers of primer/bond application with a brush and photoactivated for 20 seconds.
  Interventions: Procedure: Gingival displacement; Procedure: Enamel and dentin etched; Procedure: Wash and dry; Device: Total-etch adhesive system; Procedure: Photoactivated
- No retraction and total-etch (Active Comparator): Application of total-etch adhesive system: enamel and dentin etched with 35% phosphoric acid, wash, dry, two layers of primer/bond application with a brush and photoactivated for 20 seconds.
  Interventions: Procedure: Enamel and dentin etched; Procedure: Wash and dry; Device: Total-etch adhesive system; Procedure: Photoactivated
- Retraction and self-conditioning (Active Comparator): Gingival displacement with a gingival cord (#0, #00 or #000) prior to the restoration. Application of self-conditioning adhesive system: selective enamel etched with 35% phosphoric acid, wash, dry, one layer of acid/pirmer on enamel and dentin with a brush, one layer of bond with a brush and photoactivated for 20 seconds.
  Interventions: Procedure: Gingival displacement; Procedure: Selective enamel etched; Procedure: Wash and dry; Device: self-conditioning adhesive system; Procedure: Photoactivated
- No retraction and self-conditioning (Active Comparator): Application of self-conditioning adhesive system: selective enamel etched with 35% phosphoric acid, wash, dry, one layer of acid/pirmer on enamel and dentin with a brush, one layer of bond with a brush and photoactivated for 20 seconds.
  Interventions: Procedure: Selective enamel etched; Procedure: Wash and dry; Device: self-conditioning adhesive system; Procedure: Photoactivated

INTERVENTIONS:
Procedure: Gingival displacement — Gingival displacement with a gingival cord (#0, #00 or #000) with specific spatula.
  Arms: Retraction and self-conditioning; Retraction and total-etch
Procedure: Enamel and dentin etched — Enamel and dentin etched with 35% phosphoric acid for 30 and 15 seconds, respectively.
  Arms: No retraction and total-etch; Retraction and total-etch
Procedure: Selective enamel etched — Selective enamel etched with 35% phosphoric acid for 15 seconds.
  Arms: No retraction and self-conditioning; Retraction and self-conditioning
Procedure: Wash and dry — Wash and dry with absorbent paper.
Device: Total-etch adhesive system — Two layers of pirmer/bond on enamel and dentin with a brush.
  Arms: No retraction and total-etch; Retraction and total-etch
Device: self-conditioning adhesive system — One layer of acid/pirmer on enamel and dentin with a brush following to one layer of bond with a brush.
  Arms: No retraction and self-conditioning; Retraction and self-conditioning
Procedure: Photoactivated — Photoactivated for 20 seconds

SUMMARY:
The aim of this study is through a randomized clinical trial, double blind, splith-mouth, evaluate the retention rate of restorative protocols of Non-carious cervical lesion. The presence of gingival displacement with a retraction cord (yes or no) and the category of adhesive system (etch-and-rise and self-etching) will be evaluated. Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
Cervical wear is classified as a noncarious cervical lesion (NCCL), which is a pathological process characterized by loss of dental hard tissues near the cementoenamel junction (CEJ). The aim of this study is through a randomized clinical trial, double blind, splith-mouth, evaluate the retention rate of restorative protocols of Non-carious cervical lesion. The presence of gingival displacement with a retraction cord and the category of adhesive system will be evaluated. Two hundred and twenty teeth, with NCCL of depth greater than 1.5mm, of 55 healthy patients of both sexes will be select. The teeth will be randomly divided into 4 different groups according to the gingival displacement with retraction cord (yes or no) and adhesive system category (etch-and-rise and self-etching). Data will be collected, tabulated and submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers; both genres; presence of at least four non carious cervical lesions of similar dimensions in the same arc and opposite quadrants; good oral hygiene.

Exclusion Criteria:

* Presence of cavities, cracks or enamel fractures; extensive or unsatisfactory restorations; recent restorations involving the labial surface; dentures or orthodontics; presence of periodontal disease and,or parafunctional habits; systemic disease and, or severe psychological; constant use of analgesic and, or anti-inflammatory or allergic response to dental products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Success rate of noncarious cervical lesions restorations according to the World Dental Federation criterion | 36 mounths
  Evaluate the success rate of NCCL restoration with a 36 mounths follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soares PV, Machado AC, Zeola LF, Souza PG, Galvao AM, Montes TC, Pereira AG, Reis BR, Coleman TA, Grippo JO. Loading and composite restoration assessment of various non-carious cervical lesions morphologies - 3D finite element analysis. Aust Dent J. 2015 Sep;60(3):309-16. doi: 10.1111/adj.12233. PMID 25312697
- [Result] Grippo JO, Simring M, Coleman TA. Abfraction, abrasion, biocorrosion, and the enigma of noncarious cervical lesions: a 20-year perspective. J Esthet Restor Dent. 2012 Feb;24(1):10-23. doi: 10.1111/j.1708-8240.2011.00487.x. Epub 2011 Nov 17. PMID 22296690
- [Result] Ritter AV, Grippo JO, Coleman TA, Morgan ME. Prevalence of carious and non-carious cervical lesions in archaeological populations from North America and Europe. J Esthet Restor Dent. 2009;21(5):324-34. doi: 10.1111/j.1708-8240.2009.00285.x. PMID 19796301
- [Result] Michael JA, Townsend GC, Greenwood LF, Kaidonis JA. Abfraction: separating fact from fiction. Aust Dent J. 2009 Mar;54(1):2-8. doi: 10.1111/j.1834-7819.2008.01080.x. PMID 19228125
- [Result] Loguercio AD, Luque-Martinez I, Lisboa AH, Higashi C, Queiroz VA, Rego RO, Reis A. Influence of Isolation Method of the Operative Field on Gingival Damage, Patients' Preference, and Restoration Retention in Noncarious Cervical Lesions. Oper Dent. 2015 Nov-Dec;40(6):581-93. doi: 10.2341/14-089-C. Epub 2015 Jul 9. PMID 26158415
- [Result] Kim SY, Lee KW, Seong SR, Lee MA, Lee IB, Son HH, Kim HY, Oh MH, Cho BH. Two-year clinical effectiveness of adhesives and retention form on resin composite restorations of non-carious cervical lesions. Oper Dent. 2009 Sep-Oct;34(5):507-15. doi: 10.2341/08-006C. PMID 19830963
- [Result] Peumans M, De Munck J, Mine A, Van Meerbeek B. Clinical effectiveness of contemporary adhesives for the restoration of non-carious cervical lesions. A systematic review. Dent Mater. 2014 Oct;30(10):1089-103. doi: 10.1016/j.dental.2014.07.007. Epub 2014 Aug 3. PMID 25091726